CLINICAL TRIAL: NCT01518049
Title: Clinical Validation of the Rating Scale for Psychotic Depression (RAS-PD)
Status: Completed | Type: Observational
Sponsor: Søren Dinesen Østergaard (Other)
Responsible Party: Sponsor-Investigator, Søren Dinesen Østergaard, Principal Investigator, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: N-20110029
Record Dates: First submitted 2012-01-21; First posted 2012-01-25 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Affective Disorders, Psychotic
Keywords: Affective Disorders, Psychotic; Psychometrics; Biological Markers
MeSH Terms: conditions — Affective Disorders, Psychotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to develop a scale to measure the severity of depression with psychotic symptoms (psychotic depression). Furthermore, we hope to detect potential biomarkers (substances in the blood) which can aid in the detection of psychotic depression.

Main hypothesis: A clinically valid rating scale measuring the severity of psychotic depression can be developed.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling ICD-10 criteria DF32.3 or DF33.3
* At least 18 years old
* Legally competent
* Informed consent (oral & written)

Exclusion Criteria:

* Insufficient Danish Language skills
* Moderate to severe dementia
* Abuse of psychoactive substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inpatients or outpatients at Danish Psychiatric Hospitals fulfilling criteria for unipolar depression with psychotic symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren D Østergaard, MD, Principal Investigator — Aahus University Hospital
Locations (1):
- Unit for Psychiatric Research, Aalborg Psychiatric Hospital, Aarhus University Hospital, Aalborg, Denmark

REFERENCES:
- [Result] Ostergaard SD, Pedersen CH, Uggerby P, Munk-Jorgensen P, Rothschild AJ, Larsen JI, Gotzsche C, Sondergaard MG, Bille AG, Bolwig TG, Larsen JK, Bech P. Clinical and psychometric validation of the psychotic depression assessment scale. J Affect Disord. 2015 Mar 1;173:261-8. doi: 10.1016/j.jad.2014.11.012. Epub 2014 Nov 18. PMID 25462426